CLINICAL TRIAL: NCT06930131
Title: Effect of Anomia Rehabilitation Combined With Metacognitive Training in Patients With Chronic Vascular Aphasia
Acronym: METALEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/22/0503; 2024-A01842-45 (Other: ANSM)
Record Dates: First submitted 2025-02-19; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Aphasia; Stroke
Keywords: Aphasia; Stroke; Chronic; Cognitive rehabilitation; SCED
MeSH Terms: conditions — Aphasia; Stroke; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 6 weeks phase A (Baseline) (Other)
  Interventions: Behavioral: Semantic rehabilitation
- 7 weeks phase A (Baseline) (Other)
  Interventions: Behavioral: Semantic rehabilitation
- 8 weeks phase A (Baseline) (Other)
  Interventions: Behavioral: Semantic rehabilitation

INTERVENTIONS:
Behavioral: Semantic rehabilitation — Semantic rehabilitation, consisting of validated lexico-phonological training exercises

SUMMARY:
The postulate of this study is that rehabilitation combining linguistic and metacognitive training will result in a significant improvement in language performance correlated with changes in functional cerebral connectivity networks. In addition, it could potentiate the generalisation of effects to verbal and non-verbal communication skills, having a direct impact on patients' quality of life. This research is a prospective, randomized controlled, open-label, single-centre study. It is part of the management of patients with aphasia who have suffered a cerebral infarction and aims to evaluate the effect of combined language semantics/metacognition rehabilitation.

DETAILED DESCRIPTION:
Vascular aphasia occurs after 20 to 25% of strokes and leads to anomia or word-finding difficulties in many patients. Speech therapy, which is the standard treatment, notably employs Semantic Feature Analysis (SFA). SFA aims to teach patients a strategy that helps activate semantic links strongly associated with the target word, thereby facilitating word retrieval.

Moreover, a growing number of studies suggest combining metacognitive strategy training with language rehabilitation in brain-injured patients, particularly in reading comprehension, communication skills, and anomia, could improve cognitive and language recovery outcomes. In rehabilitation, metacognitive strategy training can be used to enhance and/or compensate for cognitive function deficits. Patients are repeatedly exposed to discrepancies between the patients performance evaluations and expectations. Findings indicate improvements in trained tasks and transfer effects to similar tasks.

While studies have examined the effects of linguistic training on one hand and the impact of metacognitive abilities on the other, to the investigators knowledge, no study has assessed the effect of a combined linguistic and metacognitive training approach in post-stroke aphasic patients on behavioral and imaging variables. This study postulates that rehabilitation combining linguistic and metacognitive training will lead to a significant improvement in language performance, correlated with changes in functional brain connectivity networks. Furthermore, it may enhance the generalization of effects to both verbal and non-verbal communication skills, directly impacting patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* First cerebral infarction
* Chronic phase (> 3 months)
* Patient affiliated to a health insurance scheme
* Usual french language
* Severity score measures using the Boston Diagnostic Aphasia Examination battery scale corresponding to the mild or moderate level (score greater than or equal to 2)

Exclusion Criteria:

* Contraindication to undergoing brain MRI
* Cognitive impairment pre-existing stroke (CQI code > 3.4) (Law et al., 1995)
* Chronic alcohol or drug abuse
* Unstabilised psychiatric illness
* Uncorrected sensory deficits
* Diagnosed as having a progressive general pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Performance at the "TD-264" untrained naming items task | Baseline, Up to 8 weeks, Up to 13 weeks
  The "TD-264 untrained naming items task" is a naming task of 264 images. Words corresponding to the images correctly named are "set success" and words wrongly named are "set treatment".
  The score at the task is composite :
  * reaction time allowing the speed of evocation to be measured will be measured with the Audacity software (https://audacity.fr/).
  * accuracy will be rated
    1. quantitatively : number of "set success"
    2. qualitatively : description of naming behaviors
  Scores are all from 0 to 264. 0 being the worst performance possible and 264 being the best performance possible.

SECONDARY OUTCOMES:
Reorganization of patients' functional connectivity maps compared to healthy volunteers | Up to 8 weeks ; Up to 13 weeks
  Reorganization of the functional connectivity of patients measured by the difference between the activation maps at the end of phase A and at the end of phase B, thanks to the acquisition of resting functional MRI sequences on the MRI dedicated to research (acquisition of resting-state MRI sequences)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No